CLINICAL TRIAL: NCT00739401
Title: Endologix Powerlink® Suprarenal Proximal Cuff
Brief Title: Suprarenal Proximal Cuff Study for Treatment of Abdominal Aortic Aneurysm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP04-002; IDE G990139 (Other: FDA)
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: AAA; Aneurysm; Suprarenal; Proximal; Cuff; Extension; Endograft; Endovascular repair; EVAR; Endoleak; Type I
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm; Endoleak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Test subjects requiring endovascular treatment of abdominal aortic or aorto-iliac aneurysms including a proximal cuff extension.
  Interventions: Device: Suprarenal Proximal Cuff Extension

INTERVENTIONS:
Device: Suprarenal Proximal Cuff Extension — Powerlink 25 and 28mm Suprarenal Proximal Extensions augmenting the 25 and 28mm Powerlink bifurcated stent graft

SUMMARY:
The use of a suprarenal extension device during the index AAA procedure to accommodate the patient's anatomy and to prevent or repair leakage.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Informed consent understood and signed
* Will comply with post-treatment follow-up requirements up to 5 years
* Candidate for Powerlink Infrarenal Bifurcated Graft

Exclusion Criteria:

* Life expectancy < 2 years
* Participating in another clinical research study
* Pregnant or lactating women
* Patient has other medical or psychiatric problems, which in the opinion of the Investigator, precludes them from participating in the Study
* Creatinine level > 1.7mg/dl
* Renal transplant patient
* Patient with > 75% renal artery stenosis and not eligible for PTA/stent intervention prior to suprarenal device fixation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-05-05 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Beasley, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; William M. Bogey, MD, Principal Investigator — East Carolina University Brody School of Medicine; Robert Feldman, MD, Principal Investigator — Munroe Regional Medical Center; Stuart Harlin, MD, Principal Investigator — Sacred Heart Hospital - Pensacola Research; Jeffrey Lawson, MD, Principal Investigator — Duke University; William Moore, MD, Principal Investigator — Lexington Medical Center; Charles Thompson, MD, Principal Investigator — Orlando Regional Medical Center; Thomas E. Topper, MD, Principal Investigator — Deaconess Hospital - The Heart Group
Locations (8):
- United States (8):
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Orlando Regional Hospital, Orlando, Florida
  - Sacred Heart Hospital - Pensacola Research Consultants, Pensacola, Florida
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Deaconess Hospital - The Heart Group, Evansville, Indiana
  - Duke University Hospital, Durham, North Carolina
  - East Carolina University - Brody School of Medicine, Greenville, North Carolina

REFERENCES:
- [Background] Parmer SS, Carpenter JP; Endologix Investigators. Endovascular aneurysm repair with suprarenal vs infrarenal fixation: a study of renal effects. J Vasc Surg. 2006 Jan;43(1):19-25. doi: 10.1016/j.jvs.2005.09.025. PMID 16414382
- [Result] Harlin SA, Beasley RE, Feldman RL, Thompson CS, Williams JB. Endovascular abdominal aortic aneurysm repair using an anatomical fixation technique and concomitant suprarenal orientation: results of a prospective, multicenter trial. Ann Vasc Surg. 2010 Oct;24(7):921-9. doi: 10.1016/j.avsg.2010.05.008. PMID 20831993
- See also: Sponsor Information — http://www.endologix.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Suprarenal Proximal Cuff Extension: Test subjects requiring endovascular treatment of abdominal aortic or aorto-iliac aneurysms including a proximal cuff extension.
  Suprarenal Proximal Cuff Extension: Powerlink 25 and 28mm Suprarenal Proximal Extensions augmenting the 25 and 28mm Powerlink bifurcated stent graft
Period: Overall Study
Arm/Group | Suprarenal Proximal Cuff Extension
Started | 44
Completed | 3
Not Completed | 41
Not completed — patients were not due for the 2 year follow-up | 34
Not completed — Death | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: All available data is reported
Arm/Group | Suprarenal Proximal Cuff Extension
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — For the purpose of this study, only Race was considered.
  Participants
    Race: White | 37
    Race: Non-White | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28 (5.5)
Ankle-Brachial Index(ABI) [Mean (Standard Deviation); unit: ratio] — The ankle-brachial pressure index or ankle-brachial index is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm. Population: All available data has been reported
  ratio
    Ankle-brachial index (ABI) - left: number analyzed (Participants) | 9
    Ankle-brachial index (ABI) - left | 1.01 (0.20)
    Ankle-brachial index (ABI) - Right: number analyzed (Participants) | 9
    Ankle-brachial index (ABI) - Right | 1.0 (0.17)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Proximal Type I Endoleak
Description: The primary study endpoint is defined as the incidence of type I proximal endoleak at 30 days post-treatment.
Time Frame: Within 30 Days
Population: Out of the 44 subjects enrolled 2 subjects withdrew even before reaching the 30day follow-up visit mark. Thus, 42 subjects were analyzed for the primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Suprarenal Proximal Cuff Extension
Number analyzed (Participants) | 42
Participants | 2

2. Secondary Outcome: Number of Subjects With Major Adverse Events
Description: All cause death, AAA rupture, Conversion / Explant, Coronary Intervention, Myocardial Infarction, Renal Failure, Respiratory Failure, Secondary Procedure, Stroke
Time Frame: Within 30 days
Population: All available data has been reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Suprarenal Proximal Cuff Extension
Number analyzed (Participants) | 44
Participants
  All-Cause Death | 0
  AAA rupture | 0
  Conversion / Explant | 0
  Coronary Intervention | 0
  Myocardial Infarction | 0
  Renal Failure | 1
  Respiratory Failure | 1
  Secondary Procedure | 0
  Stroke | 0

3. Secondary Outcome: Number of Participants With Stent Graft Integrity and Performance
Description: Number of Participants with Stent Fracture, Stent Graft Obstruction, Loss of device Integrity and Stent Migration - Core Lab reported Stent Graft Integrity Evaluation Results
Time Frame: 30 days
Population: All available data has been reported
Measure: Count of Participants; unit: Participants
Arm/Group | Suprarenal Proximal Cuff Extension
Number analyzed (Participants) | 40
Participants
  Stent Fracture | 0
  Stent Graft Obstruction | 0
  Loss of Device Integrity | 0
  Stent Graft Migration | 0

4. Secondary Outcome: Endoleak
Description: Type I (Attachment Site), Type II (Collateral), and Indeterminant type of Endoleak.
  Endoleak diagnosis results as reported by the Core Lab.
Time Frame: 30 days
Population: All available data at 30 days is reported
Measure: Count of Participants; unit: Participants
Arm/Group | Suprarenal Proximal Cuff Extension
Number analyzed (Participants) | 40
Participants
  Type I (Attachment site) | 2
  Type II (Collateral) | 6
  Indeterminant | 1

5. Secondary Outcome: Aneurysm Morphology Changes
Description: Aneurysm morphology changes (Maximum Daimeter) as reported by CoreLab.
Time Frame: 30 days
Population: All available data for 30 days has been reported
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Suprarenal Proximal Cuff Extension
Number analyzed (Participants) | 40
mm | 54 (8.7)

6. Secondary Outcome: Renal Function
Description: Renal function as measured by serum creatinine. Laboratory results,
Time Frame: 30 days
Population: All available 30 day data has been reported.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Suprarenal Proximal Cuff Extension
Number analyzed (Participants) | 37
mg/dL | 1.08 (0.35)

7. Secondary Outcome: Aneurysm Morphology Changes
Description: Aneurysm morphology changes (Volume) as reported by CoreLab.
Time Frame: 30 days
Population: All available data for 30 days has been reported
Measure: Mean (Standard Deviation); unit: cubic cm(cm^3)
Arm/Group | Suprarenal Proximal Cuff Extension
Number analyzed (Participants) | 40
cubic cm(cm^3) | 170 (56)

ADVERSE EVENTS:
Time Frame: 2 year. All Cause mortality reported through 2 years. SAEs reported through 1 year. Non SAEs reported through 2 years
Description: Specific Adverse Event terms are not collected. Events have been reported using a custom coding with organ system class. This applies to both SAEs and Non SAEs.
Arm/Group | Suprarenal Proximal Cuff Extension
All-Cause Mortality (participants affected / at risk) | 3/44
Serious Adverse Events (participants affected / at risk) | 11/44
Other Adverse Events (participants affected / at risk) | 12/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suprarenal Proximal Cuff Extension (N=44)
Blood and Lymphatic Disorders (Blood and lymphatic system disorders) | 2 (2)
Cardiac Disorders (Cardiac disorders) | 2 (3)
Gastrointestinal Disorders (Gastrointestinal disorders) | 5 (7)
Implant-Related Events (Product Issues) | 3 (4)
Musculoskeletal Disorders (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Other- SFA Rupture (Vascular disorders) | 1 (1)
Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Supplemental Procedure (Surgical and medical procedures) | 3 (3)
Vascular Disorders (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suprarenal Proximal Cuff Extension (N=44)
Blood and Lymphatic System Disorder (Blood and lymphatic system disorders) | 4 (5)
Cardiac Disorders (Cardiac disorders) | 1 (2)
Endocrine disorders (Endocrine disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
General disorders (General disorders) | 6 (9)
Infections and Infestations (Infections and infestations) | 4 (4)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (inc cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Product issues (Product Issues) | 4 (4)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 3 (4)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Surgical and medical procedures (Surgical and medical procedures) | 8 (11)
Vascular disorders (Vascular disorders) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No